CLINICAL TRIAL: NCT03322345
Title: Characterizing the Effect of Dopamine on Markers of Lymph Re-circulation in Fontan-associated Protein-losing Enteropathy
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Joshua Meisner, Pediatric Cardiology Fellow, University of Michigan
Other Study IDs: LYMPH-DOPA-PLE
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Dopamine; Protein-Losing Enteropathies; Lymphatic System; Lymph; Catecholamine; Single-ventricle; Congenital Heart Disease
Keywords: lymph flow; Fontan
MeSH Terms: conditions — Protein-Losing Enteropathies; Univentricular Heart; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Dopamine Added: Patients with protein losing enteropathy (PLE) that have an exacerbation such that their treating physicians decide to add continuous dopamine infusion to their current therapies.
- No dopamine added (control): Patients with protein losing enteropathy (PLE) that have an exacerbation such that their treating physicians decide to add new therapies to their current therapies but that do not require the addition of continuous dopamine infusion.

SUMMARY:
Patients that have undergone a Fontan procedure (surgical correction for single ventricle congenital heart disease) may develop a complication known as protein-losing enteropathy (PLE). Some studies suggest PLE is primarily caused by impaired lymph flow. Use of continuous dopamine infusion can improve PLE. Evidence suggests the effect of dopamine may be through its effect on lymphatic function. This observational study looks at markers of lymph flow and PLE symptoms after treatment using dopamine and other standard therapies during disease exacerbations.

DETAILED DESCRIPTION:
For infants and newborns who have a heart defect at birth that leaves them with one functional ventricle, there is a series of surgeries that are required to allow survival. These surgeries ultimately lead to a common heart and great blood vessel circulation called a cavopulmonary anastomosis (Fontan). This has allowed for survival into adulthood from universally fatal outcome in infancy. However, the non-physiologic blood flow patterns of the Fontan pathway do result in certain complications, including protein losing enteropathy (PLE), which occurs in 3.7-13.4% of patients. PLE is denoted by the loss of protein, fats, and other key nutrients into the intestines, which can lead to significant morbidity. Recent evidence suggests that this is in part mediated by impaired flow of lymph from the intestines, which is carried by the parallel vascular system called the lymphatic system. Lymphatics return these nutrients and the fluid that leaks out of the blood vessels throughout the body back into the blood circulatory system by functioning as a series of pumps with one-way valves. While few treatments exist from PLE, evidence demonstrates continuous infusion of dopamine can help resolve PLE symptoms. Studies of isolated lymphatic vessels demonstrate that dopamine may increase the ability of lymphatic vessels to pump harder. This suggests the mechanism of action of dopamine in PLE is increasing the return of lymph in the non-physiologic blood flow patterns of Fontan patients. However, the link between improved return of lymph and improvement in PLE has not been established. Therefore, the investigators have designed this study to test whether markers of lymphatic flow and heart pump function improve when patients start continuous dopamine therapy (a standard practice at the University of Michigan for PLE). This involves tracking markers of lymphatic recirculation through serial testing of blood and monitoring of PLE symptoms before and after the start of dopamine and other standard of care therapies. From these data, the investigators will correlate the monitored changes in lymph recirculation with changes in PLE symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Males and females with Fontan physiology of any age
* Must have protein losing enteropathy with current worsening who require additional therapies
* Participant consent or parental/guardian consent and participant assent

Exclusion Criteria:

* Patients with inflammatory bowel disease (i.e Crohn's, ulcerative colitis)
* Patients with systemic autoimmune disease (i.e. Systemic Lupus Erythematous)
* Patients with primary immunodeficiency syndromes
* Patients with nephrotic syndrome
* Patients with anemia
* Patients less than 31 pounds

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will be prospective cohort of patients who have undergone Fontan surgery and are currenty followed within the University of Michigan Congenital Heart Center. The target populations are patients with protein losing enteropathy (PLE) that are having increased disease symptoms requiring additional treatment. Those that have PLE refractory to other treatments and require the addition of continuous dopamine infusion to their treatment regimen will be recruited to the dopamine group. Those that have PLE worsening that require the addition of other treatments except the initiation of continuous dopamine infusion will be recruited to the control group.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2019-04-09 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change in CD4 counts | Baseline to 6 months
  The change in the number of circulating CD4 lymphocytes will be tracked at multiple time points from baseline to 6 months after start of additional treatment (dopamine and control)
Change in fatty acid profile | Baseline to 6 months
  The change in the relative ratios of free fatty acids absorption into the the plasma will be tracked at multiple time points from baseline to 6 months after start of additional treatment (dopamine and control)
Change in vitamin D3 | Baseline to 6 months
  The change in the levels of vitamin D3 absorbed and circulating in the plasma will be tracked at multiple time points from baseline to 6 months after start of additional treatment (dopamine and control)

SECONDARY OUTCOMES:
Change in albumin infusion requirements | Baseline to 6 months
  The change in the number of albumin infusions per month will be tracked each month from baseline to 6 months after start of additional treatment (dopamine and control)
Change in IVIG infusion requirements | Baseline to 6 months
  The change in the number of IVIG infusions per month will be tracked each mother from baseline to 6 months after start of additional treatment (dopamine and control)
Change in PLE symptoms | baseline to 6 months
  Change in symptoms of protein losing enteropathy as determined by the protein losing enteropathy assessment tool (PLEAT) at multiple time points from baseline to 6 months after initiation of additional treatment (dopamine and control)
Change in quality of life | baseline to 6 months
  Change in quantitative quality of life metrics as assessed by the Pediatric Quality of Life Inventory (PedsQL) at multiple time points from baseline to 6 months after initiation of additional treatment (dopamine and control)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Schumacher, MD, MS, Principal Investigator — University of Michigan Division of Pediatric Cardiology; Joshua Meisner, MD, PhD, Principal Investigator — University of Michigan Division of Pediatric Cardiology
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided